CLINICAL TRIAL: NCT00419575
Title: Renal Transplantation With Immune Monitoring
Status: Completed | Type: Observational
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Matthew J. Koch, Washington University
Other Study IDs: 06-0867
Record Dates: First submitted 2007-01-05; First posted 2007-01-08 (Estimated); Last update posted 2008-06-05 (Estimated); Status verified 2008-06

CONDITIONS: Renal Transplantation; Immunosuppression
Keywords: renal; transplantation; immunosuppression; monitoring

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

SUMMARY:
The aim of this observational study is to evaluate an FDA approved immune system monitoring assay (Immunknow, Cylex Inc. Columbia, MD) in renal transplant recipients using standard immunosuppression and prophylaxis protocols from the time of transplantation through a twelve month follow-up period. The primary endpoint will be the incidence of acute rejection and infection and any correlation of these events to an assay that may be a measure of recipient immune response. Secondary endpoints will include evaluation of renal function, patient and graft survival, incidence of post-transplantation lymphoproliferative disorder and duration and extent of lymphocyte depletion.

DETAILED DESCRIPTION:
As compared to previous eras, renal transplantation is a procedure associated with low acute rejection rates and excellent one year graft survival. Despite this success, long term graft survival rates have not improved significantly. The reasons for late graft loss are multi-factorial, but include chronic rejection and infection. Thus, avoidance of chronic over immunosuppression is tantamount in avoiding graft or patient threatening infection, while avoidance of under immunosuppression is necessary to prevent graft loss from acute or chronic rejection. Renal allograft loss from a particular viral pathogen, BK virus, has become evident in the era of modern immunosuppression and likely reflects relative over immunosuppression. We, and others, have used BK detection as an imprecise marker of over immunosuppression to help guide adjustments in chronic immunosuppressive therapy. While screening for the presence of BK virus is helpful in avoiding over immunosuppression and potential graft loss from BK nephropathy, a correlate assay is not readily available that provides evidence of under immunosuppression, indicating risk of graft loss from rejection.

At present, a proven assay to measure the strength of the immune system is unavailable, and the only definite markers of over or under-immunosuppression remain infection and rejection, respectively. A tool to help tailor chronic immunosuppressive therapy and decrease the incidence of either of these two extremes would be of significant value in helping to prolong allograft survival and decrease the risk of immunosuppressive therapy in renal transplant recipients.

In this observational study, we plan to use a standard immunosuppressive regimen as well as standard infection prophylaxis with the addition of an immune monitoring assay (ImmunoKnow). This assay measures ATP production by recipient T cells and has been proposed as a marker of immune function. While of interest, there are as yet, no published studies describing the utility of this test for immune monitoring in adult renal transplant recipients. As this assay remains unproven as a viable tool to define over or under immunosuppression, we will be blinded to the ImmunoKnow results during the course of the study. The results from the immune monitoring assay will only be used in a retrospective analysis to determine if there is any clinically relevant correlation between the values obtained and episodes of rejection, infection, or the development of donor specific antibodies. If a significant correlation is suggested, further evaluation in subsequent studies and eventual incorporation into prospective patient care may be warranted.

ELIGIBILITY:
Inclusion Criteria:

1. All consenting adult renal transplant recipients (age 18 years of age or older)
2. Females of childbearing age must have a negative pregnancy test performed at the time of admission for transplantation
3. Patient or guardian agrees to participate in the study and signs the informed consent.
4. Patients already consented to another study, if allowed by the study sponsor and PI of that study.

Exclusion Criteria:

1. Pregnant women or nursing mothers
2. Any patient who, in the opinion of the investigator, has a significant medical or psychosocial problem that should preclude them from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Kidney transplant recipients.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2006-10; Study Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew J Koch, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine/Barnes-Jewish Hospital, St Louis, Missouri, United States